CLINICAL TRIAL: NCT00340119
Title: Prospective Study of Inflammatory Markers and Genes as Predictors of Atherosclerotic Cardiovascular Disease in Dialysis Patients
Brief Title: Genetic Susceptibility to Cardiovascular Disease in Patients on Kidney Dialysis
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905125; 05-C-N125
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-03-01

CONDITIONS: End Stage Renal Disease; ESRD
Keywords: CHOICE Cohort; End Stage Renal Disease; Epidemiology; Prevention; Single Nucleotide Polymorphisms; ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

SUMMARY:
This study, done in collaboration with Johns Hopkins University School of Public Health in Baltimore, Maryland, will examine the role of genes in the development of atherosclerotic cardiovascular disease (CVD) in patients undergoing kidney dialysis. The rate of illness and death from CVD among patients on dialysis is extraordinarily high, accounting for about 50 percent of deaths. Blood levels of inflammatory markers are elevated in these patients, strongly predicting illness and death from CVD. The discovery of gene variants related to the inflammatory process in atherosclerotic CVD may lead to better medical treatments and improved survival in patients with end-stage kidney disease.

Participants of John's Hopkins University's CHOICE (Choices for Healthy Outcomes in Caring for End-Stage Renal Disease) program are included in this study. Blood samples previously collected from these patients will be analyzed in the laboratory for genes that might be associated with the inflammatory process and atherogenesis.

DETAILED DESCRIPTION:
Background:

The CHOICE (Choices for Healthy Outcomes in Caring for End stage renal disease) study is a national prospective cohort study of 1,041 incident dialysis patients aged 19 to 95 recruited in 81 dialysis clinics between October 1995 and June 1998, and is overseen by the Johns Hopkins University School of Public Health.

The discovery of genetic associations offers the potential to direct clinical management in order to prevent ASCVD (Atherosclerotic Cardiovascular Disease) and improve survival in patients with end stage renal disease (ESRD).

Objectives:

In Collaboration with investigators of the CHOICE cohort, we propose to assess the role of variants in genes related to the inflammatory process on atherosclerotic cardiovascular disease (ASCVD) incidence.

Eligibility:

Eligibility is independent of age, race, ethnicity, and gender. However, no participants in this cohort are less than 19 years of age.

Design:

Frozen buffy coats from 871 patients will be sent to the LGD, and DNA will be extracted.

Singles nucleotide polymorphisms (SNPs) within coding regions, upstream or downstream regulatory regions or in intronic regions of candidates genes will be genotyped.

The first candidate genes under study include IL6, IL10, TGFB1, Beta Fibrinogen, LTA, and STAT3.

Blood samples and relevant clinical data will be provided by Johns Hopkins University School of Public Health, Department of Epidemiology with only numerical code which links samples and clinical data. While Johns Hopkins University will retain patient identifier information, the LGD will have no way of identifying the person from whom the blood, subsequent DNA, and clinical data are obtained.

The samples are maintained in our repository and curated through our central Laboratory database.

Destruction or loss of clinical samples or data will be recorded in our database and cannot impact the study participants in any way.

At the completion of this protocol, we will retain the samples for future use. We understand that studies subsequent to the completion of this protocol will require additional OHSR/IRB approval prior to commencement.

ELIGIBILITY:
* INCLUSION CRITERIA:

Original eligibility criteria for enrollment in the CHOICE cohort included: 1) new onset of chronic outpatient renal replacement therapy in the last 3 months, 2) ability to give informed consent to participate in the study, 3) age 19 years or older, 4) ability to speak English or Spanish.

EXCLUSION CRITERIA:

The entire set of 871 samples available to the LGD will be analyzed. No subject will be excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 871 (Estimated)
Dates: Start 2005-03-21; Study Completion 2012-03-01

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dean, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Longenecker JC, Coresh J, Klag MJ, Levey AS, Martin AA, Fink NE, Powe NR. Validation of comorbid conditions on the end-stage renal disease medical evidence report: the CHOICE study. Choices for Healthy Outcomes in Caring for ESRD. J Am Soc Nephrol. 2000 Mar;11(3):520-529. doi: 10.1681/ASN.V113520. PMID 10703676
- [Background] Longenecker JC, Coresh J, Powe NR, Levey AS, Fink NE, Martin A, Klag MJ. Traditional cardiovascular disease risk factors in dialysis patients compared with the general population: the CHOICE Study. J Am Soc Nephrol. 2002 Jul;13(7):1918-27. doi: 10.1097/01.asn.0000019641.41496.1e. PMID 12089389
- [Background] Georges JL, Loukaci V, Poirier O, Evans A, Luc G, Arveiler D, Ruidavets JB, Cambien F, Tiret L. Interleukin-6 gene polymorphisms and susceptibility to myocardial infarction: the ECTIM study. Etude Cas-Temoin de l'Infarctus du Myocarde. J Mol Med (Berl). 2001 Jun;79(5-6):300-5. doi: 10.1007/s001090100209. PMID 11485024